CLINICAL TRIAL: NCT01695850
Title: Chinese Herbal Medicine (MaZhiRenWan) for Functional Constipation: a Prospective, Double-blinded, Double-dummy, Randomized Controlled Study
Brief Title: A Double-blinded,Double-dummy Clinical Trial of Chinese Herbal Medicine (MaZiRenWan) for Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HHSRF09101501
Record Dates: First submitted 2012-09-27; First posted 2012-09-28 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Functional Constipation; Gastrointestinal Disorders
Keywords: Randomized controlled trial; Drugs,Chinese Herbal; Constipation/drug therapy
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Sennosides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MZRW (Experimental): MZRW is composed of Fructus Cannabis (HuoMaRen), Radix et Rhizoma Rhei (DaHuang), Radix Paeoniae Alba (BaiShao), Semen Armeniacae Amarum (KuXingRen), Fructus Aurantii Immaturus (ZhiShi) and Cortex Magnoliae Officinalis (HouPo).
  Interventions: Drug: MZRW; Drug: placebo
- Senna (Active Comparator): Senna is a stimulant laxative which facilitates the passage of stools by altering intestinal electrolyte transport and increasing intestinal motor activity.
  Interventions: Drug: Senna; Drug: placebo
- Placebo (Placebo Comparator): Placebo MZRW and Placebo Senna
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MZRW — Patients are instructed to dissolve a sachet of granules (7.5g) in 150ml of hot water; they take this solution orally twice daily for 8 weeks.
  Other Names: Hemp Seed Pill
  Arms: MZRW
Drug: Senna — Patients are instructed to take 2 tablets at the bedtime for 8 weeks.
  Other Names: Senokot
  Arms: Senna
Drug: placebo — The placebo MZRW is made from dextrin (76.03%), tea essence (23.61%), gardenin (0.02%) and caramel (0.34%) to achieve color, smell, taste and texture comparable to MZRW granules.The placebo Senna is made of starch and colour to achieve comparable appearance to Senokot.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of a Chinese herbal proprietary medicine, MaZiRenWan (MZRW), by comparing with stimulant laxative western medicine (WM), senna, and placebo for patients with functional constipation (FC) in excessive TCM syndrome.

DETAILED DESCRIPTION:
Functional constipation (FC) is a common clinical complaint. Despite the effectiveness of MaZiRenWan (MZRW) for alleviating FC symptoms has been proofed in the previous study.Given the results of the dose determination study and placebo-controlled study of MZRW, we hypothesize that MZRW is more useful than senna (senokot), a commonly used WM drug for constipation, for FC patients in excessive TCM syndrome.This is a prospective, double-blind, double dummy, randomized, controlled trial. After a 2-week run-in, eligible FC patients (Rome III) in excessive TCM syndrome will randomly be assigned to CHM arm (MZRW and WM placebo), WM arm (senna and CHM placebo) or placebo arm (CHM placebo and WM placebo). Patients will undergo an 8-week treatment and an 8-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* either gender aged 18 to 65 years
* have FC diagnosed as Rome III criterial
* have diagnosis of Excessive Constipation according to the TCM theory
* complete spontaneous bowel movement (CSBM) ≦2times/w
* severity of constipation≧3pts (7 pts scale from 0 to 6pts) and the overall scoring of constipation-related symptoms≧6pts (6items in 7pts scale) for self symptom assessment in the run-in period
* normal colonic evaluation (colonoscopy or barium enema) within 12 months
* normal liver and renal function in blood test within 3 months

Exclusion Criteria:

* drug-induced constipation
* secondary causes of constipation (i.e. medical history of diabetes mellitus and thyroid disease)
* abdominal surgery (i.e. Caesarean operation)
* severe diseases (i.e. cancer and acute present asthma)
* allergy to CHM (i.e. G6PD deficiency), senna and tartrazine
* pregnancy or breast-feeding
* psychiatric or addictive disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
the responder rate for CSBM during the treatment period | 8 weeks
  a clinically meaningful endpoint by combining an objective measure (number of bowel movement) with a subjective measure (feelings of patients as to completeness of defecation,Patients with a mean increase of ≧1 complete spontaneous bowel movement(CSBM)/wk compared with the baseline(wk1-2) will be defined as responders

SECONDARY OUTCOMES:
the responder rate for CSBM during the follow-up period | 8 weeks
  Participants with a mean increase of complete spontaneous bowel movement (CSBM)>=1 movement per week compared with the last 14 days of the run-in period were defined as responders
Individual assessment of constipation and related symptoms | 18 weeks
  severity of constipation, sensation of straining, incomplete evacuation, bloating, abdominal pain / cramping, nausea, and passing of gas) was recorded using a 7-point ordinal scale (0 = not at all and 6 = very severe
the changes of colonic transit time | 18 weeks
  It is estimated by using a commercially available radio-opaque Sitzmarks capsule (Konsyl Pharmaceuticals, US). Each gelatine capsule contained 24 barium sulphate embedded polyvinyl chloride markers measuring 1mmx4.5mm. Plain radiographs of the abdomen will be obtained after the swallow of capsule for five days (120 hours) before and after 8 weeks treatment period.
Global symptom assessment | 18 weeks
  Participants were asked to rate their impression of change in constipation by comparing with their baseline (Wk2) at the visits during the treatment (Wk6), end of treatment (Wk10) and end of follow-up (Wk18) with scores from 0 to 6 represented markedly worse or better respectively. The response categories were collapsed to simply "improved" for score 4 to 6, "same" for score 3 or "worse" for score 0 to 2.
Success of blinding | 18 weeks
  the success of blinding is evaluated for both investigator and patients as to whether CHM, WM or placebo had been taken
safety profiles | 18 weeks
  Assessed by determining the important adverse events reported in the participants ' diaries, follow-up interviews,and clinical laboratory evaluationse.g., liver and renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Xiang Bian, MD, Ph. D, Principal Investigator — School of Chinese Medicine, Hong Kong Baptist University
Locations (1):
- School of Chinese Medicine, Hong Kong Baptist University, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Zhong LLD, Cheng CW, Kun W, Dai L, Hu DD, Ning ZW, Xiao HT, Lin CY, Zhao L, Huang T, Tian K, Chan KH, Lam TW, Chen XR, Wong CT, Li M, Lu AP, Wu JCY, Bian ZX. Efficacy of MaZiRenWan, a Chinese Herbal Medicine, in Patients With Functional Constipation in a Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2019 Jun;17(7):1303-1310.e18. doi: 10.1016/j.cgh.2018.04.005. Epub 2018 Apr 12. PMID 29654915
- [Derived] Zhong LL, Cheng CW, Chan Y, Chan KH, Lam TW, Chen XR, Wong CT, Wu JC, Bian ZX. Chinese herbal medicine (Ma Zi Ren Wan) for functional constipation: study protocol for a prospective, double-blinded, double-dummy, randomized controlled trial. Trials. 2013 Nov 4;14:366. doi: 10.1186/1745-6215-14-366. PMID 24180235